CLINICAL TRIAL: NCT03400267
Title: The Effect of Opioids on P2Y12 Receptor Inhibition in Patients With ST-Elevation Myocardial Infarction Who Are Pre-treated With Crushed Ticagrelor
Acronym: ON-TIME 3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: A.H. Tavenier (Other)
Collaborators: Isala (Other)
Responsible Party: Sponsor-Investigator, A.H. Tavenier, Master of Science, Isala
Organization: Isala (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ON-TIME 3
Record Dates: First submitted 2017-10-30; First posted 2018-01-17 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: STEMI; STEMI - ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Acetaminophen; Fentanyl

STUDY DESIGN:
Intervention Model Description: randomized controlled trial, with randomization to either paracetamol intravenously or fentanyl.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paracetamol (Active Comparator): Patients are randomized to paracetamol 1000 mg iv or fentanyl 1-2 mcg/kg with a maximum of 4 mcg/kg iv.
  Interventions: Drug: Paracetamol
- fentanyl (Active Comparator)
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Paracetamol — Patients are randomized to paracetamol 1000 mg iv or fentanyl 1-2 mcg/kg with a maximum of 4 mcg/kg iv.
  Arms: paracetamol
Drug: Fentanyl — Patients are randomized to paracetamol 1000 mg iv or fentanyl 1-2 mcg/kg with a maximum of 4 mcg/kg iv.
  Arms: fentanyl

SUMMARY:
Fast and accurate platelet inhibition is an important therapeutic goal in the acute treatment of patients with ST-segment elevation myocardial infarction (STEMI). Platelet inhibitory effects induced by normal oral P2Y12 receptor antagonists, for example ticagrelor, are delayed in STEMI patients undergoing primary percutaneous coronary intervention (primary PCI), which may be attributed to impaired absorption affecting drug pharmacokinetics (PK) and pharmacodynamics (PD). Another therapeutic goal in the acute treatment of STEMI is reduction of sympathetic stress and catecholamine release, thereby improving the balance between the demand for and supply of oxygen, by analgesia like fentanyl of morphine. To date, there are no studies that have specifically assessed the pharmacodynamics influences of fentanyl on platelet inhibition in STEMI patients who are pre-treated with crushed ticagrelor tablets. Therefore, In the ON-TIME-3 study, the investigators seek to show the influence of fentanyl on platelet inhibition in STEMI patients who are pre-treated with crushed ticagrelor in the ambulance.

ELIGIBILITY:
Inclusion Criteria:

i. age ≥18 years

ii. referred by ambulance paramedics to Isala (Zwolle) or Zuyderland Hospital (Heerlen)

iii. diagnosed in the ambulance with STEMI defined as:

1. ongoing chest pain >30 minutes and <12 hours duration and
2. ST-segment elevation >0.1 milliVolt in at least 2 contiguous leads

iv. ongoing chest pain with a pain score (NRS) ≥4

v. the patient has been informed of the nature of the study, agrees to its provisions and has provided verbal informed consent in the pre-hospital phase followed by written informed consent in hospital

Exclusion Criteria:

i. presenting with cardiogenic shock; defined as:

1. systolic blood pressure <90 mmHg and
2. heart rate >100/min and
3. peripheral oxygen saturation <90% (without oxygen administration)

ii. patients with a nasogastric tube in situ or requiring a nasogastric tube

iii. patients who already received fentanyl or paracetamol <2 hours prior to randomization

iv. patients on current treatment with P2Y12 inhibitors (ticagrelor, clopidogrel or prasugrel)

v. allergy to morphine or paracetamol

vi. patients with recent major bleeding complications or contraindication to dual antiplatelet therapy:

1. hypersensitivity to aspirin or ticagrelor
2. current use of (new) oral anticoagulation
3. history of bleeding diathesis or known coagulopathy
4. active bleeding
5. refusal of blood transfusions
6. history of intracerebral mass, aneurysm, arteriovenous malformation, or hemorrhagic stroke
7. known severe liver dysfunction

vii. received any organ transplant or is on a waiting list for any organ transplant

viii. patients undergoing dialysis

ix. pregnant or lactating female

x. patients currently participating in another investigational drug or device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
platelet reactivity | directly post-PCI or 1 hour post-angiography
  Platelet reactivity units (PRU) directly post-PCI or 1 hour post-angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Isala clinics, Zwolle, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided